CLINICAL TRIAL: NCT00374751
Title: Phase I/II Study of the Use of Vertebral Intracavitary Cement and Samarium (VICS) for Painful Vertebral Metastases
Brief Title: Effect of Samarium on the Relief of Pain Due to Vertebral Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Hani Ashamalla, MD, Chairman of Radiation Oncology, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYM-354
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Cancer; Metastasis; Pain
Keywords: Samarium; Kyphoplasty; Pain management; Bone metastases; Histologically proven malignancy in the primary site; Radiographic evidence of bone metastasis; Significant pain equal or more than score 5; Karnofsky Performance status >40; The patient must sign a study specific informed consent
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Pain; Agnosia | interventions — Samarium; Samarium-153

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Samarium (153SM) (Experimental): Injection of Samarium (153SM)
  Interventions: Drug: Samarium (153SM)

INTERVENTIONS:
Drug: Samarium (153SM) — The Samarium is introduced into the vertebral cavity using a 2-way valve by the radiation oncologist. The cement is then introduced via the same 2-way valve into the vertebral cavity by the neurosurgeon.

SUMMARY:
Cancer cells may spread from the primary site to the vertebrae resulting in their deformity. The standard treatment for this case is removal of the cancer deposits in the vertebra and filling the induced cavity with a cement like substance.

The investigators are studying the effects (good or bad) of adding samarium (a radioactive substance) to the cement that is injected into the induced cavity.

DETAILED DESCRIPTION:
Protocol:

1. Patients with bone metastases will be identified and discussed in the weekly joint Neuroscience meeting held in Radiation Oncology Department.
2. If the patient is eligible to this study, the protocol will be offered to him/her. If the patient accepts; informed consent will be obtained.
3. The case will be scheduled jointly by Neurosurgeon and Radiation Oncologist.
4. Radiation physicist orders the radioactive samarium.

During the procedure:

1. Neurosurgical procedure ( kyphoplasty/vertebroplasty) is performed as standard using . mild general sedation and local anesthesia.
2. Once a cavity is identified in fluoroscopy, the trocar is secured. The volume and pressure of the kyphoplasty balloon are recorded.
3. According to standard practice; only the radiation team (Radiation oncologist, Physicist) is handling the radioactive material. All work is done under sterile conditions.
4. Two mCi. of Samarium is prepared after serial dilution steps under radiation precautions in the department of radiation oncology and material is transferred to OR.
5. 0.5ml of "Head Cement" is administered first to act as a seal.
6. The Samarium is then introduced into the vertebral cavity using a 2-way valve by the Radiation Oncologist. Total of 0.5ml (Samarium+0.2ml radio opaque material)
7. The "Foot cement" (0.5 ml) is then introduced via the same 2-way valve into the vertebral cavity by the neurosurgeon to flush any remains of radioactivity in the system.
8. The two way valve is then removed and the rest of kyphoplasty/vertebroplasty is ensued as per their ordinary protocol.
9. Final volume of cement injected is recorded.
10. After securing the wound, all devices, syringes, gloves and basins used for handling the radioactive substance are collected in a "red bag" and stored by radiation safety officer in the hot lab. till full radioactive decay.
11. The room is scanned after patient's discharge, any spillage should be reported to radiation safety officer and normal procedures for environmental protection are ensued.

Post Procedure:

1. Normal neurosurgical recovery room protocol is employed. No radiation precautions needed.
2. Patient can be discharged home. No delays because of radiation precautions
3. Once patient is cleared, a nuclear imaging scan is obtained with Gamma camera. The ratio of uptake in the vertebra to background is calculated. Moreover, Full body scan is obtained to identify other areas of uptake if any.
4. A second nuclear imaging scan is done on the 4th day of the procedure (Two half Lives) to document significant decay and calculate dose.
5. MRI/CT scan of the area treated should be done in 4 weeks to assess outcome.
6. Clinical follow up is obtained at 2, 4 weeks and in 3 months. Careful pain score assessment is included in each time (Use Study Flow Sheet)

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18 years of age or older
* The patient must have histologically proven malignancy in the primary site (breast, prostate, or lung)
* The patient must have a radiographic evidence of bone metastasis, and this must have been performed within 8 weeks prior to enrollment in the study. Acceptable studies include plain radiographs, radionuclide bone scans, computed tomography scans, magnetic resonance imaging, and PET-CT scans.
* The patient must have an intact anterior wall of spinal canal
* The patient must have significant pain (score 6 or above,)which appears to be related to the radiographically documented metastatic vertebra(e) in concern, as measured by the "Visual Analog Scale"
* The patient must be surgically and medically accepted for vertebroplasty/kyphoplasty operation
* Karnofsky Performance status >40
* Expected life expectancy of 6 months or greater, as estimated by the physician in charge.
* The patient must sign a study specific informed consent prior to enrollment

Exclusion Criteria:

* Epidural soft tissue component
* Patients with vertebral metastases and with clinical or radiographic evidence of spinal cord or cauda equina impingement (effacement) or compression
* Inability to undergo anesthesia
* Hematologic primary malignancies Patients received systemic radiotherapy (89SR or 153SM)within 30 days prior to enrollmen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-05; Primary Completion 2014-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To determine the effect of intravertebral injection of Samarium on the relief of pain | 6 months
  Measuring the pain by the Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hani Ashamalla, MD, FCCP, Principal Investigator — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States